CLINICAL TRIAL: NCT01578070
Title: A Single-centre Study Evaluating the Safety of ViscoGel® and Its Safety and Efficacy as an Adjuvant in Act-HIB® Vaccine Administered by Intramuscular Injection to Healthy Volunteers in a Single-blind Randomised, Parallel-group Design
Brief Title: Single-center Study Evaluating the Safety and Efficacy of Viscogel® as Adjuvant in Act-HIB® Vaccine
Acronym: VSG-2011-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viscogel AB (Industry)
Collaborators: Karolinska Institutet (Other); Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSG-2011-101
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Other and Unspecified Vaccines and Biological Substances Causing Adverse Effects in Therapeutic Use
MeSH Terms: interventions — Hiberix; poly(ethylmethacrylate)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ViscoGel® and 0.2μg Act-HIB® (Experimental)
  Interventions: Biological: ViscoGel® and 0.2μg Act-HIB®
- 0.2μg Act-HIB® (Experimental)
  Interventions: Biological: 0.2μg Act-HIB®
- ViscoGel® and 2μg Act-HIB® (Experimental)
  Interventions: Biological: ViscoGel® and 2μg Act-HIB®
- 2μg Act-HIB® (Experimental)
  Interventions: Biological: 2μg Act-HIB®
- 10μg Act-HIB® (Active Comparator)
  Interventions: Biological: 10μg Act-HIB®

INTERVENTIONS:
Biological: 0.2μg Act-HIB® — 0.2μg Act-HIB® vaccine, IM (intramuscular) on day 0 of phase B.
  Arms: 0.2μg Act-HIB®
Biological: ViscoGel® and 0.2μg Act-HIB® — Pre-selected dose of ViscoGel® (from phase A) and Act-HIB® vaccine, IM (intramuscular) on day 0 of phase B.
  Arms: ViscoGel® and 0.2μg Act-HIB®
Biological: ViscoGel® and 2μg Act-HIB® — Pre-selected dose of ViscoGel® (from phase A) and 2μg Act-HIB® vaccine, IM (intramuscular) on day 0 of phase B.
  Arms: ViscoGel® and 2μg Act-HIB®
Biological: 2μg Act-HIB® — 2μg Act-HIB® vaccine, IM (intramuscular) on day 0 of phase B.
  Arms: 2μg Act-HIB®
Biological: 10μg Act-HIB® — Clinical standard dose of 10μg Act-HIB® vaccine, IM (intramuscular) on day 0 of phase B.
  Arms: 10μg Act-HIB®

SUMMARY:
The purpose of this study is to show that ViscoGel® is safe when administrated alone and as an adjuvant together with Act-HIB® vaccine in healthy volunteers and to evaluate the quantitative and qualitative effect on the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed a written informed consent consistent with ICH GCP guidelines and local legislations prior to participation in the trial.
* Subjects who are healthy and with no relevant medical history as determined by the investigator.
* Subject that has not previously been known to be infected with or vaccinated against HIB, or exposed to patients diseased with HIB within a 4 months period prior to screening.
* Male and non-lactating female subjects 22-50 years of age.
* Two negative pregnancy tests if female (at screening and day 0)
* Contraceptive use if female i.e. using a highly effective contraceptive method (implants, injectables, combined oral contraceptives, intra-uterine devices [including hormonal intra-uterine devices], sexual abstinence or vasectomised partner) for at least one month before dosing and willing to use it for at least one month after dosing.
* Able to read and write Swedish.

Exclusion Criteria:

* Known allergy to any component in Act-HIB, or who have had a serious reaction after previous administration of a vaccine.
* Fever or acute disease including fever.
* Receipt of immunoglobulins or blood products within three months prior to screening.
* Donation of blood or suffered of blood loss of 450 ml within 3 months (4 months if female) prior to screening.
* Donation of plasma within 14 days prior to screening.
* Participation in other clinical study within 3 months prior to screening or previously dosed in this study.
* Known or suspected immunodeficiency.
* Vaccination received within a 2 months period prior to screening.
* Any condition where regular use of inhaled, topical or oral corticosteroid is used.
* Any condition where use of immunosuppressant is needed, e.g rheumatoid arthitis, cancer, transplantation, or treatment with immunomodulators, e.g. anti-TNF alpha, methotrexte, thioguanine, cyclophosphamide, cyclosporine, tacrolimus.
* Smoker or user of other nicotine products at the discretion of the investigator.
* Drug or alcohol abuse or history of drug or alcohol abuse in the past 5 years prior to screening.
* Any medical condition or other circumstances that in the opinion of the investigator might interfere with the study.
* Abnormal clinically significant laboratory values, ECG findings, vital signs or physical examination findings as judged by the investigator.
* Inability to adhere to the protocol including plans to move from the area.
* Use of any prohibited medication (including dietary supplements and herbal medication) within 2 weeks or 7 half-lives (whichever is longer) of day 0.
* Any positive result at screening for serum hepatitis B surface antigen (HBsAG), hepatitis C antibody (anti-HCV) or human immunodeficiency virus (HIV) I and II.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence and type of adverse events, severe adverse events and SUSAR | Up to 28 days post injection
  Phase A: 3 consecutive groups each of 10 subjects. Planned dose of ViscoGel® (provided that the data safety monitoring board deemed the previous dose level to be safe): 25mg, 50mg and 75mg.

SECONDARY OUTCOMES:
Change in HIB antibody serum titer | 28 days post vaccination
  Phase B: The ViscoGel® dose administrated will be chosen after evaluation of safety and tolerance in Phase A. 2 subjects from group 1 and 2 subjects from group 3 will initially receive ViscoGel® dose (from phase A) with Act-HIB non-randomized. The remaining subjects will be randomized to 5 different treatment arms. Group 1; ViscoGel® with 0.2µg Act-HIB, Group 2; 0.2µg Act-HIB, Group 3; ViscoGel® with 2µg Act-HIB, Group 4; 2µg Act-HIB and Group 5 10µg Act-HIB is given. Blood samples are obtained at baseline and post-injection for assessment of HIB antibody serum titer.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Al-Tawil, MD/PhD, Principal Investigator — KTA
Locations (1):
- Karolinska Trial Alliance, Stockholm, Sweden

REFERENCES:
- [Derived] Neimert-Andersson T, Binnmyr J, Enoksson M, Langeback J, Zettergren L, Hallgren AC, Franzen H, Lind Enoksson S, Lafolie P, Lindberg A, Al-Tawil N, Andersson M, Singer P, Gronlund H, Gafvelin G. Evaluation of safety and efficacy as an adjuvant for the chitosan-based vaccine delivery vehicle ViscoGel in a single-blind randomised Phase I/IIa clinical trial. Vaccine. 2014 Oct 14;32(45):5967-74. doi: 10.1016/j.vaccine.2014.08.057. Epub 2014 Sep 16. PMID 25218298